CLINICAL TRIAL: NCT05259501
Title: Remote Methadone Ingestion Surveillance Trial (RMIST): A Novel and Practical Opioid Use Disorder Treatment Approach During and After the COVID-19 Pandemic
Brief Title: Remote Methadone Ingestion Surveillance Trial (RMIST)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Madhukar H. Trivedi, MD, Professor of Medicine, University of Texas Southwestern Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: CTN-0120 RMIST; STU-2023-0912; UG1DA020024 (NIH)
Record Dates: First submitted 2022-02-10; First posted 2022-02-28 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Opioid Use Disorder
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Guided video recording with tamper-evident packaging (Experimental): This method uses automated visual recognition web-based platform and QR tamper-evident labels to enhance the security of the take-home regimen currently used in methadone clinics. Single-use liquid methadone bottles are made tamper-evident through the application of a QR security label.
  Interventions: Other: RMIST

INTERVENTIONS:
Other: RMIST — RMIST will involve:
  1. A study automated visual recognition web-based platform accessible on the participant's smartphone web browser.
  2. A supply of methadone in single use bottles and previously described packaging to be kept securely at the methadone clinic/lab setting.

SUMMARY:
The Remote Methadone Ingestion Surveillance Trial (RMIST) will explore a potential method of methadone ingestion surveillance that may mitigate patient safety risks of take-home methadone treatment regimens while minimizing the risk of diversion and evaluating the acceptability and feasibility of these monitoring methods. The method utilizes an innovative existing technology.

DETAILED DESCRIPTION:
The Remote Methadone Ingestion Surveillance Trial (RMIST) aims to evaluate the performance and acceptability of a remote methadone ingestion surveillance that may mitigate the patient safety risks of take-home methadone treatment regimens for opioid use disorder (OUD) while minimizing the risk of diversion. Data describing the monitoring performance and patient acceptability of the method will inform investigators of the feasibility of using remote surveillance technology to monitor medication for OUD and mitigate treatment barriers. This study will lay the groundwork for a safe and robust remotely monitored methadone treatment platform that addresses long-standing accessibility and acceptability barriers to treatment for OUD.

ELIGIBILITY:
Inclusion Criteria:

* Be male or female, 18-65 years of age
* Currently receiving methadone maintenance treatment (MMT) for the treatment of opioid use disorder (OUD)
* Currently receiving a take-home methadone regimen of no more than three days per week (with or without COVID-19 exceptions)
* Possess an internet-connected computer or smartphone with a front facing camera.

Exclusion Criteria:

* Drug overdose requiring hospitalization within the last 12 months
* Currently or soon to be in jail or prison; currently on probation; currently in any inpatient overnight facility as required by court of law or have pending legal action or other situation that could prevent participation in the study or in any study activities
* Pregnant women
* Serious psychiatric disorders that would interfere with study participation as determined by the study site Medical Clinician
* Any participant that, according to the study team, may find it difficult to adhere to study procedures (e.g., no internet access, etc.) or are unable to operate the web-based platform for remote methadone ingestion

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2025-01-15 (Actual); Primary Completion 2025-03-13 (Actual); Study Completion 2025-03-13 (Actual)

PRIMARY OUTCOMES:
Methadone treatment adherence as measured by the number of time-stamped Medication Consumption Events (MCE) and Missed Detection Events (MDE). | Week 3
  Methadone treatment adherence as measured by the number of time-stamped Medication Consumption Events (MCE) and Missed Detection Events (MDE). i. MCEs occur any time a participant has consumed medication as detected by the web-based monitoring platform video recording. i. MDEs occur whenever a participant misses a dose during the dosing window and whenever there are user errors or platform issues. MDEs will be grouped based on commonly documented issues (e.g., platform malfunction, participant error, participant nonadherence, etc.).
Platform usability as measured by number of and self-reported reasons for occasions participants need assistance. | Weeks 1-3
  Number of occasions participants needed assistance from clinic or study staff to complete the remote monitoring process and self-reported reasons for accidental MDSs (Missed Detection Events).

OTHER OUTCOMES:
Patient-perceived advantages and disadvantages of a web-based remote methadone ingestion monitoring platform | Week 3
  Measured by survey-based assessments designed to evaluate topics related to significant barriers to receiving OUD treatments identtified by the Substance Abuse and Mental Health Services Administration (SAMHSA) - acceptability, accessibility, and privacy.

CONTACTS AND LOCATIONS:
Overall Officials: Madhukar H Trivedi, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- UNM Addiction and Substance Abuse Program, Albuquerque, New Mexico, United States

IPD SHARING:
Plan to Share IPD: Yes
This study will comply with the NIH Data Sharing Policy and Implementation Guidance (https://grants.nih.gov/grants/policy/data_sharing/data_sharing_guidance.htm). Investigators will also register and report results of the trial in ClinicalTrials.gov, consistent with the requirements of the Policy on the Dissemination of NIH-Funded Clinical Trial Information and the Clinical Trials Registration (https://grants.nih.gov/policy/clinical-trials/reporting/understanding/nih-policy.htm).
  Primary data for this study will be available to the public in the NIDA data repository, per NIDA CTN policy. For more details on data sharing please visit https://datashare.nida.nih.gov/.
  The primary outcome publication will be included along with study underlying primary data in the data share repository, and it also will be deposited in PubMed Central http://www.pubmedcentral.nih.gov/ per NIH Policy (http://publicaccess.nih.gov/).
Time Frame: Immediately following publication. No end date
Access Criteria: Anyone who wishes to access the data
URL: https://datashare.nida.nih.gov/

DOCUMENTS (1):
  • Informed Consent Form (2024-12-04): https://cdn.clinicaltrials.gov/large-docs/01/NCT05259501/ICF_000.pdf